CLINICAL TRIAL: NCT01219933
Title: An Open-label, Single-arm Study to Describe Glucocorticoid Use in Rheumatoid Arthritis Patients Treated With Tocilizumab in Daily Clinical Practice and to Evaluate Systematic Glucocorticoid Dose Reduction Once Low Disease Activity is Reached (ACT-ALONE)
Brief Title: A Study of Glucocorticoid Use to Evaluate Systematic Methylprednisolone Reduction in Patients With Rheumatoid Arthritis on Background RoActemra/Actemra (Tocilizumab) (ACT-ALONE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25252; 2010-019694-15
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methylprednisolone; tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methylprednisolone; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: methylprednisolone — starting dose >/= 1 mg and </= 20 mg orally daily, according to dose-reduction schedule
Drug: tocilizumab [RoActemra/Actemra] — background therapy: 8 mg/kg iv every 4 weeks

SUMMARY:
This open-label, single-arm study will assess the use of glucocorticoids (GC) in daily clinical practice and will evaluate the dose reduction of glucocorticoids once low disease activity is achieved in patients with rheumatoid arthritis tre ated with GC and background RoActemra/Actemra (tocilizumab) 8mg/kg intravenously every 4 weeks. In the non-interventional phase, the use of GC in daily clinical Belgian practice will be evaluated and described. This period of maximum 6 mont hs will allow those patients to obtain the inclusion criteria for the secondary interventional phase. In the interventional phase, a systematic GC dose reductio n schedule will be evaluated in patients having achieved low disease activity wh ile receiving the same background therapy with RoActemra/Actemra 8 mg/kg. Methyl prednisolone will be given from a starting dose of >/= 1 mg to </=20 mg orally d aily and will be tapered down. The anticipated study duration is up to 13 months

ELIGIBILITY:
Inclusion Criteria:

Non-interventional phase

* Adult patients, >/=18 years of age
* Moderate to severe active rheumatoid arthritis defined as Disease Activity Score using 28-joint count (DAS28) >/=5.1
* Patients with inadequate clinical response to a current treatment with 2 or more non-biologic disease-modifying anti-rheumatic drugs (DMARDs), one of them being methotrexate (MTX) optimally administered during a period of more than 3 months or inadequate response to a current anti-TNF therapy
* Current use of oral glucocorticoids started at least 4 weeks prior to enrolment Interventional phase
* Patients enrolled in the non-interventional phase
* Patients with low disease activity defined as DAS28 </=3.2 at Visit 2
* Use of oral glucocorticoids with methylprednisolone equivalent dose of >/=1mg and </=20mg/day at Visit 2

Exclusion Criteria:

Non-interventional & interventional phase

* Rheumatic autoimmune disease other than rheumatoid arthritis, or significant systemic involvement secondary to rheumatoid arthritis
* Functional class IV as defined by the American College of Rheumatology (ACR) Classification of Functional Status in rheumatoid arthritis
* Prior history or current inflammatory joint disease other than rheumatoid arthritis (e.g. gout)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- Belgium (15):
  - Aalst
  - Bruges
  - Brussels
  - Charleroi
  - Edegem
  - Genk
  - Gilly
  - Godinne
  - Haine-Saint-Paul
  - Heusy
  - Kortrijk
  - La Louvière
  - Liège
  - Ostend
  - Wilrijk

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenously (IV) once every 4 weeks and methotrexate (MTX) 7.5 to 25 mg per week (mg/week; per investigator's discretion, or without MTX if intolerant) for up to 13 months. Participants also received an oral glucocorticoid (GC; no product/dose limitation) until low disease activity (LDA; defined as Disease Activity Score Based on 28-Joint Count and C-reactive protein [DAS28-CRP] less than or equal to [≤]3.2), up to a maximum of 6 months. Once LDA achieved, GC was switched to methylprednisolone (MP) tablets, by mouth (PO). MP dose determined by recalculating original GC dose to obtain an equivalent MP dose (had to be greater than or equal to [≥]1 mg and ≤20 mg per day [mg/day]), which was administered for 4 weeks. If LDA continued after 4 weeks, MP dose was reduced over the following 6 months per protocol-defined dose reduction schedule to reach 0 mg within 6 months for a maximum duration of 7 months of MP treatment
Period: Overall Study
Arm/Group | Tocilizumab
Started | 68
Completed | 30
Not Completed | 38
Not completed — Adverse Event | 8
Not completed — No LDA reached | 5
Not completed — No LDA maintained | 7
Not completed — Lost to Follow-up | 3
Not completed — GC free | 1
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 8
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety observational (obs): all participants included in the study who were eligible for the study at Visit (V) 1.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg IV once every 4 weeks and MTX 7.5 to 25 mg/week per investigator's discretion, or without MTX if intolerant) for up to 13 months. Participants also received GC (no product/dose limitation) until LDA (defined as DAS28-CRP ≤3.2), up to a maximum of 6 months. Once LDA achieved, GC was switched to MP tablets, PO. MP dose determined by recalculating original GC dose to obtain an equivalent MP dose (had to be ≥1 mg and ≤20 mg/day), which was administered for 4 weeks. If LDA continued after 4 weeks, MP dose was reduced over the following 6 months per protocol-defined dose reduction schedule to reach 0 mg within 6 months for a maximum duration of 7 months of MP treatment.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Median GC Dose Taken During the Noninterventional Phase
Description: During the noninterventional phase of the study participants received GC as prescribed by the physician. Doses of all GC administered are expressed as MP equivalents.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety obs population; n (number) equals (=) number of participants analyzed for a given parameter at a specified timepoint
Measure: Median (Full Range); unit: mg
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
mg
  Start dose V1 (n=68) | 6 [2 to 40]
  Start dose (V1) for Interventional phase (n=50) | 6 [2 to 32]
  Stop dose (V2; n=50) | 4 [1 to 16]
  Change from start to stop (n=50) | 0 [-24 to 2]
  Cumulative dose from V1 to V2 (n=45) | 320 [58 to 2688]

2. Primary Outcome: Number of Participants With GC Switches During the Noninterventional Phase
Description: During the noninterventional phase of the study, once LDA was achieved, GC was switched to MP tablets.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety obs population; n=number of participants analyzed for a given parameter at a specified timepoint
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
participants | 0

3. Secondary Outcome: Percentage of Participants Able to Acheive LDA Assessed Using DAS28 While Receiving Oral GC on Background Tocilizumab Treatment During the Noninterventional Phase
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the CRP and Patient's Global Assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 ≤3.2 and oral GC intake with MP equivalent dose of ≥1 mg and ≤20 mg/day= LDA.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants | 72.1

4. Secondary Outcome: Percentage of Participants Acheiving Remission Assessed Using DAS28 While Receiving Oral GC on Background TocilizumabTreatment During the Noninterventional Phase
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the CRP and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 <2.6 = remission.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
percentage of participants | 41.2

5. Secondary Outcome: Percentage of Participants With Erosions During the NonInterventional Phase
Description: In RA, the presence, number and size of bone erosions and the number of joints with erosions on conventional radiographs (CRs) are hallmarks for diagnosis, staging and prediction of damage progression and are used for treatment monitoring in randomized controlled studies.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 57
percentage of participants
  V1 (n=57) | 47.4
  Between V1 and V2 (n=36) | 41.7

6. Secondary Outcome: Number of Erosions During the NonInterventional Phase
Description: In RA, the presence, number, and size of bone erosions and the number of joints with erosions on CRs are hallmarks for diagnosis, staging and prediction of damage progression and are used for treatment monitoring in randomized controlled studies.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: erosions
Arm/Group | Tocilizumab
Number analyzed (Participants) | 11
erosions
  V1 (n=11) | 5.1 (6.0)
  Between V1 and V2 (n=6) | 3.2 (2.3)

7. Secondary Outcome: Percentage of Participants Positive for Rheumatoid Factor (RF) During the Noninterventional Phase
Description: RF is the auto antibody directed against immunoglobulin G (IgG) and its concentration is observed in human serum or plasma. RF value higher than 20 units per milliliter (U/mL) is considered positive.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 39
percentage of participants
  V1 (n=39) | 56.4
  Between V1 and V2 (n=21) | 52.4

8. Secondary Outcome: Percentage of Participants Positive for Anti-cyclic Citrullinated Peptide (Anti-CCP) Antibody During the Noninterventional Phase
Description: Anti-CCP antibodies are important markers of bone erosion in RA. Anti-CCP antibodies were classified as positive if >7 U/mL.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 20
percentage of participants
  V1 (n=20) | 75.0
  Between V1 and V2 (n=6) | 83.3

9. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) During the Noninterventional Phase
Description: HAQ-DI is a self-reported, valid assessment of functional disability in RA. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ-DI score range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation. Timepoint was V2, or before V2 for participants withdrawn before V2.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 66
units on a scale
  V1 (n=66) | 1.7 (0.6)
  V2 (n=61) | 1.2 (0.7)
  Change from V1 to V2 (n=60) | -0.5 (0.6)

10. Secondary Outcome: DAS28-CRP During the Noninterventional Phase
Description: DAS28-CRP was calculated from the swollen joint count (SJC) and tender joint count (TJC) using the 28-joint count and CRP (mg/L). Total score range: 0 to 10, higher score indicated more disease activity. DAS28-CRP ≤3.2=LDA and >3.2 to 5.1=moderate to high disease activity, and DAS28-CRP <2.6=remission. Timepoint was V2, or before V2 for participants withdrawn before V2; DAS28-CRP values indicated in the Case Report Form (CRF) were recalculated by the data manager. The recalculated values were used in the statistical analyses.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 67
units on a scale
  V1 (n=67) | 5.4 (1.0)
  V2 (n=66) | 2.9 (1.1)
  Change from V1 to V2 (n=65) | -2.5 (1.3)

11. Secondary Outcome: DAS28-ESR During the Noninterventional Phase
Description: DAS28-ESR was calculated from the SJC and TJC using the 28 joints count and ESR (millimeters per hour [mm/hr]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-ESR ≤3.2=LDA and >3.2 to 5.1=moderate to high disease activity, and DAS28-ESR <2.6=remission. Timepoint was V2, or before V2 for participants withdrawn before V2; DAS28-ESR values indicated in the CRF were recalculated by the data manager. The recalculated values were used in the statistical analyses.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 62
units on a scale
  V1 (n=62) | 5.8 (1.0)
  V2 (n=52) | 3.3 (1.4)
  Change from V1 to V2 (n=50) | -2.7 (1.3)

12. Secondary Outcome: Clinical Disease Activity Index (CDAI) During the Noninterventional Phase
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and Physician Global Assessment (PGA) of disease assessed on 0-100 mm Visual analog scale (VAS); higher scores=greater affection due to disease activity. CDAI total score=0-76. CDAI ≤2.8=disease remission, >2.8 to 10=LDA, >10 to 22=moderate disease activity, and >22=high disease activity.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 62
units on a scale
  V1 (n=62) | 33.8 (12.2)
  V2 (n=52) | 14.6 (10.3)
  Change from V1 to V2 (n=50) | -20.4 (13.7)

13. Secondary Outcome: Median Time Interval Between V1 and V2
Description: The noninterventional phase was planned to last for a maximum of 6 months per participant. The time between V1 and V2 was measured in months.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population
Measure: Median (Full Range); unit: months
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
months | 2.3 [0.8 to 5.9]

14. Secondary Outcome: Median Dose of Tocilizumab During the Noninterventional Phase
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
mg/kg | 8.0 [8.0 to 8.0]

15. Secondary Outcome: Number of Participants With Changes in Tocilizumab Dose During the Noninterventional Phase
Description: The dose of tocilizumab could have been reduced from the recommended 8 mg/kg to 4 mg/kg in participants in the case of adverse events.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 68
participants | 1

16. Secondary Outcome: Percentage of Participants With Changes in RA Treatment During the Noninterventional Phase
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety Obs Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 66
percentage of participants | 15.2

17. Secondary Outcome: Percentage of Participants Able to Start the GC Reduction Phase at V3
Description: All participants who maintained LDA (defined as DAS28-CRP ≤3.2) from V2 to V3 were included in the interventional phase for reduction of GC.
Time Frame: V3 (7 months)
Population: Safety Int (intervention) run-in: all participants eligible to enter the interventional phase at V2 and who had taken at least 1 dose of MP.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percentage of participants | 87.8 [75.2 to 95.4]

18. Secondary Outcome: Percentage of Participants Able to Reduce Oral GCs by ≥50 Percent (%) During the Interventional Phase by V9
Time Frame: V9 (24 weeks after V3)
Population: Safety Int run-in; only those participants who completed the study at V9 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 30
percentage of participants | 93.3 [77.9 to 99.2]

19. Secondary Outcome: Percentage of Participants Able to Discontinue GCs During the Interventional Phase by V9
Time Frame: V9 (24 weeks after V3)
Population: Safety Int run-in; pnly those participants who completed the study at V9 were included in analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 30
percentage of participants | 3.3 [0.1 to 17.2]

20. Secondary Outcome: Time-Averaged GC Dose Changes During the Interventional Phase
Description: Area Under the Curve (AUC) of GC dose during the interventional phase was determined using the trapezoidal method and was calculated as:
  AUC = sigma(Ti+1 - Ti) x [(Di+1+Di)/2]
  With Di=dosage at time Ti
  It corresponds to the total GC dose received between Baseline (visit 3) and visit 9 and has been calculated only for the 30 patients achieving visit 9.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; only participants who completed the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tocilizumab
Number analyzed (Participants) | 30
mg | 341.8 (364.2)

21. Secondary Outcome: DAS28-CRP During the Interventional Phase
Description: DAS28-CRP was calculated from the SJC and TJC using the 28-joint count and CRP (mg/L). Total score range: 0 to 10, higher score indicated more disease activity. DAS28-CRP) ≤3.2=LDA and >3.2 to 5.1=moderate to high disease activity, and DAS28-CRP <2.6=remission. DAS28-CRP values indicated in the CRF were recalculated by the data manager. The cumulative DAS28 (CRP) value (AUC method) was performed using the calculated DAS28. The recalculated values were used in the statistical analyses.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 42
units on a scale
  V3 (n=42) | 2.2 (0.7)
  CV (n=27) | 2.3 (0.8)
  Change from V3 to CV (n=27) | 0.2 (0.8)

22. Secondary Outcome: HAQ-DI During the Interventional Phase
Description: HAQ-DI is a self-reported, valid assessment of functional disability in RA. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ-DI score range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation. V3, CV, and the change from V3 to CV was determined.
Time Frame: Visit 3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Obs Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
units on a scale
  V3 (n=41) | 1.0 (0.7)
  CV (n=28) | 0.8 (0.7)
  Change from V3 to CV (n=26) | 0.0 (0.4)

23. Secondary Outcome: VAS-Physician's Global Assessment of Disease Activity (GDA) During the Interventional Phase
Description: Physician's were asked to determine the overall GDA for each participant using a 100-mm VAS, where 0=no disease activity and 100=maximum disease activity. The physician marked the line corresponding to their assessment and the distance from the left edge was measured. V3, CV, and the change from V3 to CV was determined.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint. Only participants with values at both visits were included in the analysis.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 40
mm
  V3 (n=40) | 16.6 (12.5)
  CV (n=28) | 16.7 (15.9)
  Change from V3 to CV (n=26) | 3.1 (15.4)

24. Secondary Outcome: VAS for Pain (VAS-Pain) During the Interventional Phase
Description: Participants were asked to mark the line corresponding to the intensity of their pain on a 100-mm VAS, where 0=no pain and 100=worst possible pain. The distance from the left edge was measured. Change = V3 mean minus CV mean.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 43
mm
  V3 (n=43) | 19.9 (16.5)
  CV (n=28) | 24.9 (19.0)
  Change from V3 to CV (n=28) | 6.9 (22.4)

25. Secondary Outcome: SJC and TJC During the Interventional Phase
Description: TJC and SJC were assessed for 28 joints. An assessment of 28 joints for swelling and tenderness was made. Joints were assessed and classified as swollen (1)/not swollen (0) and tender (1)/not tender (0) by pressure and joint manipulation on physical examination for a total score range of 0-28. Higher scores indicated greater disease activity (tenderness/swelling). V3, CV, and the change from V3 to CV was determined.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 43
joints
  SJC V3 (n=43) | 0.9 (1.3)
  SJC CV (n=29) | 0.4 (0.9)
  SJC Change from V3 to CV (n=29) | -0.3 (0.8)
  TJC V3 (n=43) | 0.9 (1.2)
  TJC CV (n=29) | 1.8 (2.7)
  TJC Change from V3 to CV (n=29) | 1.0 (2.6)

26. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score During the Interventional Phase
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-F score for a total possible score of 0 (worse score) to 52 (better score). V3, CV, and the change from V3 to CV was determined.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 37
units on a scale
  V3 (n=37) | 37.5 (9.9)
  CV (n=26) | 35.6 (10.8)
  Change from V3 to CV (n=22) | 8.8 (19.0)

27. Primary Outcome: Type of GC Taken at the End of the Noninterventional Phase
Description: During the noninterventional phase of the study participants received GC as prescribed by the physician.
Time Frame: V1 and V2 (up to 6 months after V1)
Population: Safety obs population; n=number of participants analyzed for a given parameter at a specified timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
percentage of participants
  MP | 70.0
  Prednisolone | 28.0
  Prednisone | 2.0

28. Primary Outcome: Percentage of Participants in the Interventional Phase Who Achieved LDA and Discontinued Oral GC Within 20 Weeks
Description: The percentage of participants with rheumatoid arthritis (RA) with LDA was defined as DAS28 ≤3.2, able to discontinue oral GC within 20 weeks and at the latest at V8, confirmed at the Consolidation Visit without loss of clinical response defined as DAS28 (CRP) >3.2.
Time Frame: Visits 3 (7 months), 4 (8 months), 5 (9 months), 6 (10 months), 7 (11 months), and 8 (12 months)
Population: Intent-to-Treat (ITT) population: all participants included in the interventional GC reduction phase of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 43
percentage of participants | 58.1 [42.1 to 73.0]

29. Secondary Outcome: Short-Form 36 (SF-36) Mental Component Score (MCS) and Physical Component Score (PCS) During the Interventional Phase
Description: 36-Item Short-Form Health Survey (SF-36) is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component scores (PCS and MCS). Total of 11 variables were analyzed (8 subscales, 2 composite subscales and Question 2 "how would you rate your health in general now?" (range 1= better, 5= worst). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Higher scores reflect higher quality of life. V3, CV, and the change from V3 to CV was determined.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 37
units on a scale
  MCS V3 (n=37) | 47.0 (9.9)
  MCS CV (n=26) | 46.2 (9.0)
  MCS: Change from V3 to CV (n=22) | -4.4 (10.6)
  PCS V3 (n=36) | 42.5 (7.6)
  PCS CV (n=26) | 41.8 (8.8)
  PCS: Change from V3 to CV (n=22) | -2.1 (6.4)

30. Secondary Outcome: SF-36 Subscale Scores During the Interventional Phase
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects can also be summarized as physical and mental component scores (PCS and MCS). Total of 11 variables were analyzed (8 subscales, 2 composite subscales and Question 2 "how would you rate your health in general now?" (range 1= better, 5= worst). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Higher scores reflect higher quality of life. V3, CV, and the change from V3 to CV was determined.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 37
units on a scale
  Physical functioning V3 (n=36) | 41.52 (10.37)
  Physical functioning CV (n=26) | 41.92 (10.44)
  Change in physical functioning V3 to CV (n=22) | -1.80 (6.77)
  Physical sub-score V3 (n=37) | 40.61 (7.53)
  Physical sub-score CV (n=26) | 39.85 (8.23)
  Change in physical sub-score V3 to CV (n=22) | -2.79 (7.68)
  Bodily pain V3 (n=37) | 45.88 (8.35)
  Bodily pain CV (n=26) | 44.65 (9.70)
  Change in bodily pain V3 to CV (n=22) | -3.21 (8.67)
  General health V3 (n=37) | 43.11 (9.42)
  General health CV (n=26) | 40.82 (8.77)
  Change in general health V3 to CV (n=22) | -3.78 (7.35)
  Vitality V3 (n=37) | 50.51 (8.74)
  Vitality CV (n=26) | 48.91 (9.13)
  Change in vitality V3 to CV (n=22) | -4.37 (9.98)
  Social functioning V3 (n=37) | 45.42 (9.63)
  Social functioning CV (n=26) | 45.58 (9.29)
  Change in social functioning V3 to CV (n=22) | -2.73 (9.63)
  Emotional sub-score V3 (n=37) | 40.59 (9.98)
  Emotional sub-score CV (n=26) | 40.37 (10.53)
  Change in emotional sub-score V3 to CV (n=22) | -2.45 (10.29)
  Mental health V3 (n=37) | 47.14 (10.00)
  Mental health CV (n=26) | 45.94 (10.37)
  Change in Mental health V3 to CV (n=22) | -5.47 (10.98)

31. Secondary Outcome: CDAI Score During the Interventional Phase
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-100 mm VAS; higher scores=greater affection due to disease activity. CDAI total score=0-76. CDAI ≤2.8=disease remission, >2.8 to 10=LDA, >10 to 22=moderate disease activity, and >22=high disease activity. V3, CV, and the change from V3 to CV was determined.
Time Frame: V3 (7 months) and CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 40
units on a scale
  V3 (n=40) | 5.6 (3.8)
  CV (n=27) | 6.5 (5.4)
  Change from V3 to CV (n=25) | 1.4 (5.2)

32. Secondary Outcome: Percentage of Participants With LDA or Remission During the Interventional Phase Assessed Using CDAI
Description: The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PtGA and PGA assessed on 0-100 mm VAS; higher scores=greater affection due to disease activity. CDAI total score=0-76. CDAI ≤2.8=disease remission and >2.8 to 10=LDA.
Time Frame: Visits 3 (7 months), 4 (8 months), 5 (9 months), 6 (10 months), 7 (11 months), 8 (12 months), and 9 (24 weeks after V3) or CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 41
percentage of participants
  V3 LDA (n=40) | 85.0
  V3 Remission (n=40) | 27.5
  V4 LDA (n=41) | 82.9
  V4 Remission (n=41) | 39.0
  V5 LDA (n=38) | 81.6
  V5 Remission (n=38) | 47.4
  V6 LDA (n=35) | 71.4
  V6 Remission (n=35) | 37.1
  V7 LDA (n=33) | 75.8
  V7 Remission (n=33) | 33.3
  V8 LDA (n=31) | 80.6
  V8 Remission (n=31) | 38.7
  V9 LDA (n=29) | 69.0
  V9 Remission (n=29) | 31.0
  CV LDA (n=27) | 77.8
  CV Remission (n=27) | 33.3

33. Secondary Outcome: Percentage of Participants With LDA or Remission During the Interventional Phase Assessed Using DAS28-CRP
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joint count, the CRP and PtGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28-CRP ≤3.2 and oral GC intake with MP equivalent dose of ≥1 mg and ≤20 mg/day=LDA; DAS28 <2.6 = remission.
Time Frame: Visits 3 (7 months), 4 (8 months), 5 (9 months), 6 (10 months), 7 (11 months), 8 (12 months), 9 (24 weeks after V3) or CV (4 weeks after GC-free status, maximum of 24 weeks after V3)
Population: Safety Int run-in; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 42
percentage of participants
  V3 LDA (n=42) | 90.5
  V3 Remission (n=42) | 73.8
  V4 LDA (n=41) | 85.4
  V4 Remission (n=41) | 73.2
  V5 LDA (n=35) | 88.6
  V5 Remission (n=35) | 71.4
  V6 LDA (n=35) | 82.9
  V6 Remission (n=35) | 62.9
  V7 LDA (n=33) | 90.9
  V7 Remission (n=33) | 57.6
  V8 LDA (n=32) | 87.5
  V8 Remission (n=32) | 62.5
  V9 LDA (n=30) | 73.3
  V9 Remission (n=30) | 56.7
  CV LDA (n=27) | 88.9
  CV Remission (n=27) | 59.3

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the study from V1, 6 months before Interventional phase to CV
Groups:
- Noninterventional Phase: Participants received tocilizumab 8 mg/kg IV once every 4 weeks and MTX 7.5 to 25 mg/week according to local standard of care and at the investigator's discretion (or without MTX if intolerant) for up to 13 months. Participants also received GC (no product/dose limitation) until LDA (defined as DAS28-CRP ≤3.2), up to a maximum of 6 months.
- Interventional Phase: All participants who maintained LDA from V2 to V3 were included in the interventional phase for reduction of GC. Once LDA achieved, GC was switched to MP tablets, PO. MP dose determined by recalculating original GC dose to obtain an equivalent MP dose (had to be ≥1 mg and ≤20 mg/day), which was administered for 4 weeks. If LDA continued after 4 weeks, MP dose was reduced over the following 6 months per protocol-defined dose reduction schedule to reach 0 mg within 6 months for a maximum duration of 7 months of MP treatment.
Arm/Group | Noninterventional Phase | Interventional Phase
Serious Adverse Events (participants affected / at risk) | 4/68 | 1/43
Other Adverse Events (participants affected / at risk) | 36/68 | 26/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Noninterventional Phase (N=68) | Interventional Phase (N=43)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Attempted to commit suicide (Psychiatric disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Noninterventional Phase (N=68) | Interventional Phase (N=43)
Bronchitis (Infections and infestations) | 6 | 3
Fatigue (General disorders) | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Oedema peripheral (General disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Otosalpingitis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Body tinea (Infections and infestations) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Presyncope (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Hip surgery (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 1
Rheumatoid vasculitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.